CLINICAL TRIAL: NCT06173882
Title: The Therapeutic Effect and Standardization of Moxibustion in the Treatment of Allergic Rhinitis
Brief Title: Moxibustion Reduces Symptoms and Improves Quality of Life in Patients With Allergic Rhinitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCM for AR
Record Dates: First submitted 2023-12-05; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; moxibustion; body surface temperature
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ordinary moxibustion volume group (Placebo Comparator)
  Interventions: Behavioral: Ordinary moxibustion volume group
- First group of heavy moxibustion (Experimental)
  Interventions: Behavioral: First group of heavy moxibustion
- Second groups of heavy moxibustion (Experimental)
  Interventions: Behavioral: Second groups of heavy moxibustion

INTERVENTIONS:
Behavioral: Ordinary moxibustion volume group — Moxibustion for 10 minutes per acupoint
  Arms: Ordinary moxibustion volume group
Behavioral: First group of heavy moxibustion — Moxibustion for 20 minutes per acupoint
  Arms: First group of heavy moxibustion
Behavioral: Second groups of heavy moxibustion — Moxibustion for 30 minutes per acupoint
  Arms: Second groups of heavy moxibustion

SUMMARY:
The objective of this randomized controlled clinical trial is to compare the therapeutic effect of moxibustion on allergic rhinitis. The main questions it aims to answer are:

Based on randomized controlled trials, verify the effectiveness of moxibustion in treating allergic rhinitis Based on a real-time monitoring system for human surface temperature, discuss the differences in therapeutic effects of different moxibustion doses on allergic rhinitis

DETAILED DESCRIPTION:
Allergic rhinitis has a high incidence and is difficult to cure, seriously affecting the quality of life of patients Compare the effects of different moxibustion durations on the clinical efficacy and body surface temperature of patients with allergic rhinitis, and preliminarily explore the impact of different moxibustion doses on the efficacy of heavy moxibustion treatment for allergic rhinitis, providing evidence-based basis for clinical practice.

ELIGIBILITY:
Inclusion criteria

* Those who meet the diagnostic criteria of Chinese and Western medicine for AR;
* Age range from 18 to 75 years old, regardless of gender;
* Patients and their families are informed and agree to the study.

Exclusion criteria

* Those who are undergoing other traditional Chinese medicine external treatment methods;
* Those who have taken traditional Chinese medicine recently or during treatment;
* Individuals who are allergic to heavy moxibustion smoke and dust;
* Individuals with concomitant bronchial asthma or other respiratory system diseases;
* Patients with severe skin diseases or ulcers in the local area where moxibustion is applied;
* Pregnant and lactating patients;
* Patients with severe diseases of important organs such as the heart, liver, lungs, and kidneys;
* Those who are unable to receive treatment according to regulations due to inconvenience in work, study, transportation, or personal activities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Rhinitis VAS Visual Analog Scale（AR-VAS） | Change from baseline VAS scores at week 0(before treatment)，4 and 12.
  VAS will be used to evaluate the relief of rhinitis symptoms, with a total score of 0-10. The higher the score, the more severe the symptoms will be
Total nasal symptom scores（TNSS） | Change from baseline TNSS scores at week 0(before treatment)，4 and 12.
  The main symptoms of allergic rhinitis, the higher the score, the worse the condition

SECONDARY OUTCOMES:
Total non nasal symptom scores（TNNSS） | Change from baseline TNNSS scores at week0(before treatment)，4 and 12.
  The nasal accompanying symptoms of allergic rhinitis, qualitative evaluation of the severity of the disease, with some indicating severity and none indicating milder severity
Rhino-conjunctivitis Quality of Life Questionnaire （RQLQ） | Change from baseline RQLQ scores at week0(before treatment)，4 and 12.
  RQLQ consists of 28 items, including daily life (1-3), sleep (4-6), non nasal eye symptoms (7-13), life problems (14-16), nasal symptoms (17-20), eye symptoms (21-24), and emotions (25-28). In the 7-point system, 1 point is the best and 7 points are the worst.
Detection of serum IgE and IL-33 levels | Week0(before treatment), week 4（after treatment）.
  Immunoglobulin IgE and serum inflammatory cytokine IL-33 levels

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xie, MD, Study Director — Henan University of Traditonal Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, China